CLINICAL TRIAL: NCT02504567
Title: Laser Ablation Study for trEatment of atRial Fibrillation (LASER)
Acronym: LASER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: CardioFocus (Industry)
Responsible Party: Principal Investigator, Josep Lluis Mont Girbau, MD Phd, Hospital Clinic of Barcelona
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Laser
Record Dates: First submitted 2015-07-15; First posted 2015-07-22 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-08

CONDITIONS: Atrial Fibrillation
Keywords: Catheter Ablation; Radiofrequency; Laser; Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Laser Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laser ablation (Other): Ablation with laser catheter
  Interventions: Device: Laser ablation
- RF ablation (Other): Ablation with RF catheter
  Interventions: Device: RF ablation

INTERVENTIONS:
Device: Laser ablation — Pulmonary vein isolation using the laser ablation catheter
  Arms: Laser ablation
Device: RF ablation — Pulmonary vein isolation using the RF ablation catheter
  Arms: RF ablation

SUMMARY:
This protocol aims at assessing the efficacy of performing catheter ablation for atrial fibrillation (AF) with laser catheters versus performing it with radiofrequency (RF) catheters. In order to study laser catheter ablation efficacy, MRI analysis of the lesions 3 months after the procedure will be performed in both groups. MRI analysis will detect ablation gaps in the lesions encircling pulmonary veins. The primary endpoint will compare the number of gaps in the laser catheter and the RF group. The secondary endpoint of the study is recurrence of AF after 12 months. The target population of the study is patients with paroxysmal or persistent AF undergoing AF ablation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical recurrent AF, refractary or intolerant to at least 1 antiarrhythmic drub who are scheduled to undergo ablation of pulmonary veins (PV)
* Signed consent form.

Exclusion Criteria:

* Being under 18 years old
* Any contraindication for ablation procedure
* Impossibility to acquire DE-MRI because of contraindication (e.g. severely impaired renal function) or patient unwillingness

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-07; Primary Completion 2016-11 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Presence of large gaps in the delayed enhancement MRI (DE-MRI) | 3 months
  The presence of MRI ablation gaps around the pulmonary veins evaluated with MRI images of the patient acquired three months after the ablation procedure. A large gap is described as a GAP that is larger or equal than 20% of the vein perimeter.

SECONDARY OUTCOMES:
To determine the number of patients that present atrial fibrillation after the ablation procedure | 1 year
  The number of patients that present a recurrence in their atrial fibrillation after the ablation procedure during the first year.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, Catalonia, Spain